CLINICAL TRIAL: NCT06573515
Title: Effectiveness of High Tone Power Therapy Versus Interferential Current Therapy in Mothers With Breastfeeding-Related Neck Pain
Brief Title: High Tone Power Therapy Versus Interferential Current Therapy in Mothers With Breastfeeding-Related Neck Pain
Acronym: BFRNP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, heba Haridy, lecturer of basic science department, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0001111
Record Dates: First submitted 2024-08-13; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Breastfeeding
Keywords: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-tone power therapy group (Experimental): fifteen female patients will receive high-tone power therapy with conventional physical therapy modalities in the form of (ultrasound, massage, stretching, and strengthening exercises) 2 sessions per week for 6 weeks
  Interventions: Device: high tone power therapy
- interferential current therapy group (Experimental): fifteen female patients will receive interferential current therapy with conventional physical therapy modalities in the form of (ultrasound, massage, stretching, and strengthening exercises) 2 sessions per week for 6 weeks
  Interventions: Device: interferential current therapy
- conventional physical therapy group (Experimental): fifteen female patients will receive conventional physical therapy modalities only in the form of (ultrasound, massage, stretching, and strengthening exercises) 2 sessions per week for 6 weeks
  Interventions: Device: conventional physical therapy

INTERVENTIONS:
Device: high tone power therapy — female patients will receive high-tone power therapy using a device (HiTop 191 Medizintechnik, Rimbach, Germany) duration 30 minutes at 2 sessions per week for 6 weeks
  Arms: high-tone power therapy group
Device: interferential current therapy — female patients will receive interferential current therapy using Enraf-Nonius (ENDOMED 484, Germany)The electrode pairs will placed at a distance of at least 2.5 cm from each other. The utilized parameters will have a base frequency of 4,000 Hz, a modulation frequency range of 10 Hz-20 Hz, spectrum mode triangular, and slope 1/1 in a quadripolar manner with a beat frequency of 80 Hz. duration of treatment session 20 minutes 2 sessions per week for 6 weeks
  Arms: interferential current therapy group
Device: conventional physical therapy — female patients will receive conventional physical therapy modalities in the form of (ultrasound, massage, stretching, and strengthening exercises) 2 sessions per week for 6 weeks
  Arms: conventional physical therapy group

SUMMARY:
Breastfeeding is very essential for the growth and development of an infant. World Health Organization recommends exclusive breastfeeding of the baby for the first six months. Duration of breastfeeding ranges from 15-20 minutes and is done after every 2-3 hours. The frequency of breastfeeding is approximately 8-12 times a day. So collectively 5-6 hours in an entire day are spent while feeding the baby. Breastfeeding mothers encounter various musculoskeletal problems. These problems arise due to the inappropriate positions acquired during breastfeeding the baby. Since these positions are maintained for longer durations, they can lead to long-term postural deformities by altering the normal curvature of spine. Moreover hormonal changes of pregnancy may last from 12 weeks postpartum to 6 months postpartum. All these changes will have a long-lasting effect while performing activities of daily living, hampering baby care and self-care (Dandekar et al., 2022). In addition to breast soreness, engorgement, maternal illness, blocked ducts, and mastitis, breastfeeding-related neck pain has a high prevalence among nursing women. It is commonly associated with the adoption of awkward postures during feeding sessions. One of the most common awkward positions adopted by nursing mothers is unsupported head/neck posture, resulting in sustained neck flexion to monitor the infant during feeding. Such a sustained awkward position with excessive repetition usually puts stress on the neck and back muscles

DETAILED DESCRIPTION:
High tone power therapy is a new application with unique characteristics of electrotherapy and its main effects for the body are entering energy into the body to revitalize the body to affect and stimulate cells and inducing a resonance effect that makes vibration or an oscillation in the tissues and cells to relieve pain, enhance metabolism and distributing the pain mediators and inflammation, waste substances and nutrients; thus normalizing the cell and organizing metabolism and nerve regeneration The application of the high tone power therapy proved to be a very effective treatment that improved the extent of cervical spine mobility with significant pain alleviation in patients with cervical pain Interferential current therapy is a safe physical therapy method that has been used for many years in the treatment of musculoskeletal system disorders. It has analgesic, anti-inflammatory, sympatholytic, local vasodilatory, and muscle stimulatory actions. It shows significant analgesic effects in patients with neck pain

ELIGIBILITY:
Inclusion Criteria:

* All mothers are medically stable.
* All mothers are primiparous and currently breastfeed their infants.
* All mothers will be exclusive breastfeeding mothers.
* Their ages will be 18-35 years old.
* Their body mass index will be 18.5 to 24.9 kg/m2.
* All mothers will provide an informed consent form agreeing to participate and publication of the study results.

Exclusion Criteria:

* Mothers who were pregnant and nursing with known orthopedic and neurological conditions of the spine, upper limbs and shoulder regions prior to breastfeeding.
* Mothers had cesarean delivery.
* Mothers with cerebrovascular problems, or any disorder affect the goal of the study.
* Mothers with preterm babies, low-birth weight babies, intrauterine growth restriction, with chronic diseases like cancer, human immuno-deficiency virus (HIV), tuberculosis and with postpartum complications like postpartum hemorrhage and eclampsia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 6 weeks
  The visual analogue scale, a calibrated scale on which the patients could indicate their assessment along a 10 cm line, describes the subjective pain level. It is marked from 0 to 10, with 0 representing no pain and 10 standing for unbearable pain
Neck disability index | 6 weeks
  The Neck disability index will assess functional restriction for all patients before and after the treatment. The Neck disability index will developed to measure self-perceived disability from neck pain.
  It is a 10-item scaled questionnaire entitled the neck disability index, each item will recorded out of five for a maximum total score of 50 and a higher score indicates more patient-rated disability
Cervical range of motion device | 6 weeks
  The cervical range of motion device is made of an unbreakable polyester material; it has a comfortable frame that adjusts to the patient's head is secured with Velcro straps and has three planes. The sagittal plane meter measures flexion and extension, while the lateral plane meter measures lateral flexion; both are fluid-damped inclinometers and work by the force of gravity as the position of the head changes. The magnetic plane meter measures rotational movement in conjugation with a magnetic yoke

CONTACTS AND LOCATIONS:
Locations (1):
- Heba, Cairo, Egypt